CLINICAL TRIAL: NCT00367640
Title: Randomised,Double-blind,Placebo-controlled,Multinational,Multi-centre,Phase IIb/III Study of the Efficacy and Safety of Three Doses of Sublingual Immunotherapy (SLIT) Administered as Tablets Once Daily to Patients Suffering From Grass Pollen Rhinoconjunctivitis
Brief Title: Safety and Efficacy of Sublingual Immunotherapy (SLIT) Tablets in Grass Pollen Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO34.04
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Allergy
Keywords: Sublingual immunotherapy; Grass pollen tablet; Allergic rhinoconjunctivitis
MeSH Terms: conditions — Hypersensitivity | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 100 IR (Experimental): 100 IR grass pollen allergen extract tablet
  Interventions: Drug: 100 IR grass pollen allergen extract tablet
- 300 IR (Experimental): 300 IR grass pollen allergen extract tablet
  Interventions: Drug: 300 IR grass pollen allergen extract tablet
- 500 IR (Experimental): 500 IR grass pollen allergen extract tablet
  Interventions: Drug: 500 IR grass pollen allergen extract tablet
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: 100 IR grass pollen allergen extract tablet — One sublingual tablet daily during 4 months before pollen season and during pollen season
  Other Names: Sublingual immunotherapy tablet
  Arms: 100 IR
Drug: 300 IR grass pollen allergen extract tablet — One sublingual tablet daily during 4 months before pollen season and during pollen season
  Other Names: Sublingual immunotherapy tablet
  Arms: 300 IR
Drug: 500 IR grass pollen allergen extract tablet — One sublingual tablet daily during 4 months before pollen season and during pollen season
  Other Names: Sublingual immunotherapy tablet
  Arms: 500 IR
Drug: Placebo tablet — One sublingual tablet daily during 4 months before pollen season and during pollen season
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of SLIT compared with placebo for reduction of symptoms and rescue medication usage

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Grass-pollen related allergic rhinoconjunctivitis for at least the last 2 pollen seasons.
* Sensitised to grass pollen (positive SPT and RAST level of at least class 2).
* Total symptom score of the RRTSS during the previous pollen season greater than or equal to 12.
* Safety laboratory resuts within the references ranges

Exclusion Criteria:

* Pregnancy, breast-feeding/lactation
* Had received desensitisation treatment for grass pollen
* Treatment by immunotherapy with another allergen within the previous 5 years
* Usual contraindications of immunotherapy such as serious immunopathologic conditions or malignancies
* Treated with beta-blockers or under continuous corticotherapy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 628 (Actual)
Dates: Start 2004-11; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain DIDIER, Professor, Principal Investigator — Hôpital Rangueil-Larrey, Toulouse, France

REFERENCES:
- [Result] Didier A, Malling HJ, Worm M, Horak F, Jager S, Montagut A, Andre C, de Beaumont O, Melac M. Optimal dose, efficacy, and safety of once-daily sublingual immunotherapy with a 5-grass pollen tablet for seasonal allergic rhinitis. J Allergy Clin Immunol. 2007 Dec;120(6):1338-45. doi: 10.1016/j.jaci.2007.07.046. Epub 2007 Nov 1. PMID 17935764

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 30 NOV 2004, Last Patient Last Visit 05 SEP 2005
Period: Overall Study
Arm/Group | 100 IR | 300 IR | 500 IR | Placebo
Started | 157 | 155 | 160 | 156
Completed | 139 | 133 | 141 | 146
Not Completed | 18 | 22 | 19 | 10
Not completed — Adverse Event | 3 | 6 | 8 | 0
Not completed — Withdrawal by Subject | 8 | 11 | 8 | 6
Not completed — Any other reason not above-mentioned | 7 | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all patients who received at least one dose of investigational product and had a Retrospective Rhinoconjunctivitis Total Symptom Score (RRTSS) and at least one Rhinoconjunctivitis Total Symptom Score (RTSS) in the pollen period while on treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 IR | 300 IR | 500 IR | Placebo | Total
Number analyzed (Participants) | 142 | 136 | 143 | 148 | 569
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (6.90) | 28.7 (7.34) | 30.4 (7.45) | 29.1 (7.60) | 29.4 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 62 | 54 | 60 | 245
  Male | 73 | 74 | 89 | 88 | 324

OUTCOME MEASURES:

1. Primary Outcome: Average Rhinoconjunctivitis Total Symptom Score
Description: Average Rhinoconjunctivitis Total Symptom Score during the pollen period while participant on treatment.
  Participants assessed daily, during the pollen period, 6 rhinoconjunctivitis symptoms (sneezing, rhinorrhea, nasal pruritus, nasal congestion, ocular pruritus and watery eyes) each symptom is scored as follows: 0: no symptoms, 1: mild symptoms, 2: moderate symptoms, 3: severe symptoms. The sum of the 6 symptoms is the Rhinoconjunctivitis Total Symptom Score (RTSS) (range 0-18). The lower the score, the better the outcome.
Time Frame: Pollen period (average of 32 days in the ITT set)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale (range: 0 to 18)
Arm/Group | 100 IR | 300 IR | 500 IR | Placebo
Number analyzed (Participants) | 142 | 136 | 143 | 148
Units on a scale (range: 0 to 18) | 4.72 (3.141) | 3.58 (2.976) | 3.74 (3.142) | 4.93 (3.229)
Statistical Analysis 1: Comparison: 500 IR vs Placebo; A step-down approach is performed to address the multiplicity issue; Test type: Superiority or Other; p = 0.0006, ANCOVA — ANCOVA of the average RTSS, with treatment and pooled sites as factors, and retrospective RTSS, asthma and sensitised status as covariates
Statistical Analysis 2: Comparison: 300 IR vs Placebo; A step-down approach is performed to address the multiplicity issue; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 100 IR vs Placebo; A step-down approach is performed to address the multiplicity issue; Test type: Superiority or Other; p = 0.4606, ANCOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 4 months before the pollen period until the end of pollen period.
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse event that started on or after the first dose of the investigational product.
  Note: Serious Adverse Events and Other Adverse Events are described in Results Publication.
Arm/Group | 500 IR | 300 IR | 100 IR | Placebo
Serious Adverse Events (participants affected / at risk) | 3/160 | 1/155 | 0/157 | 0/156
Other Adverse Events (participants affected / at risk) | 74/160 | 70/155 | 76/157 | 36/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 500 IR (N=160) | 300 IR (N=155) | 100 IR (N=157) | Placebo (N=156)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 500 IR (N=160) | 300 IR (N=155) | 100 IR (N=157) | Placebo (N=156)
ORAL PRURITUS (Gastrointestinal disorders) | 41 | 40 | 31 | 8
OEDEMA MOUTH (Gastrointestinal disorders) | 10 | 7 | 5 | 0
TONGUE OEDEMA (Gastrointestinal disorders) | 9 | 4 | 5 | 0
HEADACHE (Nervous system disorders) | 14 | 22 | 23 | 21
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 23 | 14 | 18 | 5
NASOPHARYNGITIS (Infections and infestations) | 12 | 13 | 16 | 11
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 3 | 10 | 1
EAR PRURITUS (Ear and labyrinth disorders) | 7 | 5 | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No